CLINICAL TRIAL: NCT02064673
Title: Randomized Trial of Adjuvant Curcumin After Prostatectomy
Brief Title: Adjuvant Curcumin to Assess Recurrence Free Survival in Patients Who Have Had a Radical Prostatectomy
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: yair lotan (Other)
Responsible Party: Sponsor-Investigator, yair lotan, PROFESSOR, University of Texas Southwestern Medical Center
Organization: University of Texas Southwestern Medical Center (Other)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: STU 042013-080
Record Dates: First submitted 2014-02-10; First posted 2014-02-17 (Estimated); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: Prostate Cancer
Keywords: prostate cancer; radical prostatectomy
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Curcumin; Sugars

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | US Export: No

ARMS (2):
- Curcumin (Active Comparator): Curcumin 500 mg orally twice a day
  Interventions: Drug: Curcumin; Drug: placebo
- sugar pill (Placebo Comparator): placebo orally twice a day
  Interventions: Drug: Curcumin; Drug: placebo

INTERVENTIONS:
Drug: Curcumin — Curcumin or placebo 500mg by mouth twice a day for 6 months
  Other Names: Bio-Curcumin(BCM-95CG); Tumeric
Drug: placebo — placebo orally twice a day
  Other Names: sugar pill

SUMMARY:
This is a prospective study to determine if the adjuvant use of Curcumin improves recurrence-free survival.

DETAILED DESCRIPTION:
This is a prospective study to determine if the adjuvant use of Curcumin improves recurrence-free survival in patients after radical prostatectomy compared to placebo

ELIGIBILITY:
Inclusion Criteria:

* Status post radical prostatectomy for histologically confirmed adenocarcinoma of the prostate
* pathologically confirmed T1-T3 disease
* no sign of lymph node or metastatic disease
* pT1-pT3pNxMx patients in whom standard NCCN or AUA guidelines would suggest are at low risk for pelvic lymph node or metastatic disease and who would not require confirmatory imaging for metastatic disease. This includes patients with Gleason 6 or 7(T2 disease) and PSA less than 20.
* Eastern Cooperative Oncology Group(ECOG) status 0-2
* adequate renal and liver function as well as bone marrow reserve (measured serum creatinine <2mg/dl, bilirubin ≤ 1.5 mg/dl, ANC ≥ 1.5 x 10 (3) uL, platelets ≥ 50 x K/uLL, and hemoglobin ≥ 10 g/dL)
* 30-80 y/o at time of diagnosis with a life expectancy of >= 3 yrs
* focally positive surgical margins are permitted
* no plan to receive adjuvant hormone or radiation therapy
* PSA at the time of enrollment must be undetectable
* life expectancy of 3 years

Exclusion Criteria:

* must not have exceeded 3 months from time of surgery to enrollment into study
* T3b or T4 or node positive disease
* macroscopic residual disease after surgery
* hormone therapy before surgery
* history of gallbladder problems or gallstones, or biliary obstruction, unless patient had cholecystectomy
* radiation therapy as primary treatment after surgery
* INR value greater than 1.5
* AST/ALT are equal or greater than 2 times the upper limit of normal
* antiplatelet or anticoagulant agents- patients taking 81mg of Aspirin will be allowed with close observation
* history of gastric or duodenal ulcers or untreated hyperacidity syndromes
* patients who are currently taking curcumin and are unwilling to stop or plan to take curcumin during the study

Ages: 30 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 608 (Estimated)
Dates: Start 2014-05; Primary Completion 2028-06 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Serum prostate specific antigen | 3 years
  Recurrence free survival defined as a total serum prostate specific antigen of <0.2ng/ml.

CONTACTS AND LOCATIONS:
Overall Officials: Yair Lotan, MD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- UT Southwestern Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No